CLINICAL TRIAL: NCT02022800
Title: Prospective Study on Oncologic Cerebral Imagery Contribution by 18F-FDOPA Position Emission Tomography (PET) in a Multidisciplinary Meeting Therapeutic Proposal When Caring for Patients Diagnosed Primary or Secondary Cerebral Tumors
Brief Title: Prospective Study on Oncologic Cerebral Imagery Contribution by 18F-FDOPA Position Emission Tomography (PET)
Acronym: IMOTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012/56
Record Dates: First submitted 2013-11-19; First posted 2013-12-30 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2015-11

CONDITIONS: Glioma; Cerebral Metastases
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET 18FDOPA (Other): PET 18FDOPA
  Interventions: Other: PET 18FDOPA

INTERVENTIONS:
Other: PET 18FDOPA — contribution of PET 18FDOPAimagery in high level glioma diagnosis

SUMMARY:
In standard care for patients diagnosed with a primary or secondary (metastasis) cerebral tumor, there is currently complex clinical situations in which the clinic and Magnetic Resonance Imagery (MRI) do not allow for the medical team to arrive at a conclusive diagnosis. The therapeutic proposition requires then a delay in additional follow-up of at least 3 months in order to clarify the situation, with a potential delay in diagnosis and therefore therapeutic care. The contribution of cerebral molecular imagery could allow for new additional information to be brought in or to increase the confidence index in the diagnosis in order to comfort the therapeutic collective attitude proposed in the multidisciplinary meeting (MM).

3.4-dihydroxy-6-18F-fluoro-L-phenylalanine (18F-FD0PA), dopamine precursor amino-acid, Position Emission Tomography (PET), allows for the studying in vivo of the proteic transmembrane transport in gliomatous tissue; active transport happens through a sodic-independent canal, increased in malicious transformations, and in which kinetics can give an indication regarding the development of the primary tumor.

In MRIs, tumor tissue growth after injecting the contrast product translates to a rupture in the Blood-Brain Barrier (BBB), while tumor extraction from the radiopharmaceutical is independent of the state of integrity of the BBB and whose only function is metabolic tissue activity. This method of imagery thus appears as a promising contribution to conventional imagery.

Furthermore, different to 18F-FDG (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose), similar to the largely used glucose in oncologic molecular imagery, exploration of harmful glioma in 18F-FDOPA, is not compromised by background noise activity, and is almost useless in a healthy cerebral cortex, with the exception of striatal physiological fixation used as a level of reference. The best performances in terms of positive and negative predictive value were defined in the literature with a tumor/striatum threshold of 1.

According to the latest and current European recommendations, turning to PET when caring for high-level gliomas patients can be proposed in the evaluation of therapeutic responses. However, very few studies have evaluated the in-practice current clinical contributions of PET and put it into perspective with classic clinical radiological data.

DETAILED DESCRIPTION:
The primary hypothesis rests on the fact that 18F-FDOPA PET imagery can modify decisions regarding the treatment of patients during oncologic neurological MDM. It's a matter of measuring the frequency in attitude and situations changes in which these changes most often occur.

Secondly, the study will have the objective, during patient follow-up, to evaluate the pertinence of these changes in decisions, as well as the usage of PET in relation to clinical situations:

* The differential diagnosis between radionecrosis or pseudo-progression and recurrence before newly appeared contrast zones in patients diagnosed a high glioma level or metastasis and treated by radiotherapy; either with or without chemotherapy.
* The evaluation at the end of treatment with introductory level temozolomide (TMZ) (6th cycle) after adjuvant radio-chemotherapy of a high-level primary cerebral tumor.
* The evaluation of the response under anti-angeogenic treatment

The expected benefit of this study is an improvement in the patient's care. Indeed, the additional information provided by Position Emission Tomography (PET) could allow for healthcare professionals to more precociously test for recurrence and thus diminish the delay in therapeutic care. Conversely, the PET could allow for healthcare professionals to avoid over-treatment of patients for whom the MRI would wrongly indicate a recurrence. Furthermore, imagery by PET should bring a new level of additional information allowing for an increase in the confidence index when being diagnosed, thus comforting the collective therapeutic attitude proposed in the MM.

ELIGIBILITY:
Inclusion Criteria:

Patients with a historically proven high level of glimoa or of cerebral metastases

Patients who have their files presented in a neurological oncologic CMM in one of the following situations:

* Diagnosis doubt between radionecrosis and tumor progression
* Evaluation at the end of the radio and chemotherapy period
* Evaluation under anti-angiogenic 18 years or older Patients who have been informed and have signed the consent form indicated in the study Patients with insurance coverage

Exclusion Criteria:

Patients for whom having an MRI or a PET 18F-FDOPA would be contraindicated in light of any co-morbidities or allergies that it reveals

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-11; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
confidence level in the therapeutic decision regarding the results from PET 18F-FDOPA imagery, in comparison with MRI alone. | 1 year up to 2 years

SECONDARY OUTCOMES:
Validation of the decision taken with knowledge of the results from the PET 18F-FDOPA for post-operated patients | 1 year up to 2 years
evaluation of PET 18F-FDOPA contribution according to clinical situations | 1 year up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jacques DARCOURT, phd, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France

REFERENCES:
- See also: Related Info — http://www.centreantoinelacassagne.org